CLINICAL TRIAL: NCT04504162
Title: Iatrogenic Addiction to Sedation in Shanghai
Brief Title: Monitoring and Risk Prediction of Iatrogenic Sedative Hypnotics Addiction in a Shanghai Psychiatric Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: HFJiang-005
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Hypnotics and Sedatives; Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- outpatient: Patients visiting a psychiatric hospital

SUMMARY:
This study will establish a sedative and hypnotics iatrogenic addiction risk monitoring network composed of 4 psychiatric hospitals in Shanghai through standardized data construction of outpatient prescription data and personnel training. Develop a sedative-hypnotic addiction risk prediction tool based on patient prescription data, and use independent in-operation outpatient prescription data for verification, and carry out clinical application promotion.

DETAILED DESCRIPTION:
This study is a longitudinal analysis of the outpatient prescription data of psychiatric hospitals. It includes two aspects: 1) Develop evaluation methods for the risk of sedative-hypnotic addiction in psychiatric hospitals; 2) Construct a predictive model for the risk of iatrogenic addiction to sedative-hypnotics.

Step 1. Export all sedative hypnotic prescription information from the outpatient medical record system of Shanghai Psychiatric Hospital.

The data range is from January 1, 2019 to December 31, 2020. The data items that need to be exported include: patient identification information, gender, age, diagnosis, prescription drug name, drug use method, total dose, time , and the physician number of the prescription. Generate a unique patient number based on identification information (such as ID number), and merge all prescription information and electronic medical records of the same patient during the study period.

Step 2. Identify patients at risk of addiction to sedative hypnotics. This study defines the risk of addiction to sedatives and hypnotics when the outpatients appear "double off-label prescriptions". The standard of "double off-label prescriptions" is: the highest daily average dose of prescriptions obtained by patients>60 mg diazepam equivalent milligrams, and the number of consecutive prescription days>120 days. Firstly, mark whether the patient has a prescription that exceeds the specification range (over indication, over daily dose range, over treatment course) during the study period. Secondly, the analysis data set is further converted and labeled, including: all benzodiazepine doses are converted into diazepam equivalents according to the "Benzazepine Dose Conversion Table". Calculate the "average daily prescription dose" for each patient: add up the prescriptions of benzodiazepines to get the total prescription, and divide by the number of days to get the average daily prescription dose. Finally, calculate the monthly or annual cases or proportion of "double off-label prescriptions" patients who are at risk of addiction to sedatives and hypnotics.

Step 3.Establish a risk prediction model for iatrogenic addiction to sedative and hypnotics in psychiatric hospitals.

Use correlation analysis or machine learning methods to explore the formation trajectory of the "double off-label" pattern of sedative hypnotic prescriptions, and build a predictive model that can predict the formation of the "double off-label" pattern. Use a subset of prescription data to identify patients with status of "double off-label", then evaluate and review them to confirm the addiction status of sedatives and hypnotics. Use the validation subset to verify and improve the addiction risk prediction model based on the training data set.

ELIGIBILITY:
This study is a data analysis based on outpatient visit records. The research object is the prescription data of outpatient visits during the research period, that is, the prescription information of any patient visiting the outpatient clinic during the research period will be included in the analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient visiting the outpatient clinic of Shanghai mental health center during the research period will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Outpatient's prescription | Data from January 1, 2019 to December 31, 2020
  The research object is the outpatient prescription information of each independent year (2019, 2020) of each hospital (4 hospitals), including: patient identification information, gender, age, diagnosis, prescription drug name, drug use method, total dose, time , And the physician number of the prescription. Generate a unique patient number based on identification information (such as ID number), and merge all prescription information and electronic medical records of the same patient during the study period. And mark whether the patient has a prescription that exceeds the specification range (over indication, over daily dose range, over treatment course) during the study period.

IPD SHARING:
Plan to Share IPD: Undecided
Will share results within the scope of Chinese laws and regulations.